CLINICAL TRIAL: NCT04090190
Title: Inflammation in Women With Urgency Urinary Incontinence Treated With Anticholinergics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Vatche Arakel Minassian, Chief, Division of Urogynecology. Associate Professor, Harvard Medical Schoo, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000980
Record Dates: First submitted 2019-08-21; First posted 2019-09-16 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Urinary Incontinence; Urgency Urinary
Keywords: Urinary Incontinence; Urgency Urinary; Anticholinergic Treatment; Urinary Microbiome
MeSH Terms: conditions — Urinary Incontinence | interventions — oxybutynin; Solifenacin Succinate; Tolterodine Tartrate; trospium chloride; fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- standard of care anticholinergic treatment (Other): Women presenting to the Urogynecology clinic with urgency urinary incontinence symptoms will receive standard of care anticholinergic treatment and will have their urinary microbiome evaluated before and after treatment
  Interventions: Drug: Oxybutynin, Solifenacin, Tolterodine, Trospium, or Fesoterodine

INTERVENTIONS:
Drug: Oxybutynin, Solifenacin, Tolterodine, Trospium, or Fesoterodine — Study participants will be evaluated for urgency urinary incontinence and will be offered treatment with a standard of care anticholinergic medication for 6 weeks. All study participants will fill out the UDI-6 and two day bladder diary at baseline before starting anticholinergic medication treatment. Participants will then provide a urine sample and blood draw to be assessed for urinary microbiome and inflammation. Anticholinergic medication will be taken daily for 6 weeks and the same procedures (UDI-6 questionnaire, bladder diary, urine sample except the blood draw for assessment) will be performed at the 6-week time period.
  Other Names: Ditropan; Vesicare; Detrol; Sanctura; Toviaz

SUMMARY:
Urinary incontinence (UI) is a very common condition affecting women of all ages. The objective of this pilot study is to better understand the urinary microbiome and associated inflammatory markers in blood and urine in women with urgency UI. The study will assess how inflammation may affect response to standard of care anticholinergic medication treatment for urgency urinary incontinence.

DETAILED DESCRIPTION:
This study is designed as a prospective pilot study of women presenting to the Urogynecology clinic with urgency urinary incontinence symptoms who are offered treatment with a standard of care anticholinergic medication for six weeks. The patient will be asked to provide a catheterized urine sample at baseline and 6 weeks and blood draw only at baseline. Study participants will fill out a Urinary Distress Inventory-6 (UDI-6) questionnaire at baseline and fill a bladder diary for 48 hours before starting the anticholinergic medication.

The urine will be assessed by standard and enhanced urine cultures and DNA amplification and 16S rRNA sequencing for urinary microbiome along with inflammatory markers in the urine. Inflammatory markers in both the blood and urine will be measured using immunoenzyme assays.

Measurements for microbiome will be repeated for all patients at 6 weeks. Baseline urinary symptoms at enrollment and variation of symptoms after 6 weeks of anticholinergic treatment will be assessed using the UDI-6 questionnaire and a bladder diary.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (Age ≥ 50) women with Urgency Urinary Incontinence (UUI)
* English speaking
* Willing to take anticholinergics for at least 6 weeks
* Willing to complete UDI-6 and voiding diary at baseline and 6 weeks
* Willing to give urine and blood for study at baseline and 6 weeks

Exclusion Criteria:

* Have taken anticholinergic medication within the last month
* Have taken antibiotics within the last month
* Urinary Tract Infection (UTI) in the last three months
* Neurological disease (eg. Parkinson's disease, Multiple Sclerosis, etc.)
* Immunological deficiencies
* History of sexually transmitted disease (STD)
* Lack of consent
* Not ambulatory (e.g. uses a wheelchair)

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vatche Minassian, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molinuevo B, Batista-Miranda JE. Under the tip of the iceberg: psychological factors in incontinence. Neurourol Urodyn. 2012 Jun;31(5):669-71. doi: 10.1002/nau.21216. Epub 2012 Mar 30. PMID 22473905
- [Background] Hu TW, Wagner TH, Bentkover JD, Leblanc K, Zhou SZ, Hunt T. Costs of urinary incontinence and overactive bladder in the United States: a comparative study. Urology. 2004 Mar;63(3):461-5. doi: 10.1016/j.urology.2003.10.037. PMID 15028438
- [Background] Cho I, Blaser MJ. The human microbiome: at the interface of health and disease. Nat Rev Genet. 2012 Mar 13;13(4):260-70. doi: 10.1038/nrg3182. PMID 22411464
- [Background] Hilt EE, McKinley K, Pearce MM, Rosenfeld AB, Zilliox MJ, Mueller ER, Brubaker L, Gai X, Wolfe AJ, Schreckenberger PC. Urine is not sterile: use of enhanced urine culture techniques to detect resident bacterial flora in the adult female bladder. J Clin Microbiol. 2014 Mar;52(3):871-6. doi: 10.1128/JCM.02876-13. Epub 2013 Dec 26. PMID 24371246
- [Background] Thomas-White KJ, Kliethermes S, Rickey L, Lukacz ES, Richter HE, Moalli P, Zimmern P, Norton P, Kusek JW, Wolfe AJ, Brubaker L; National Institute of Diabetes and Digestive and Kidney Diseases Urinary Incontinence Treatment Network. Evaluation of the urinary microbiota of women with uncomplicated stress urinary incontinence. Am J Obstet Gynecol. 2017 Jan;216(1):55.e1-55.e16. doi: 10.1016/j.ajog.2016.07.049. Epub 2016 Aug 4. PMID 27498309
- [Background] Pearce MM, Zilliox MJ, Rosenfeld AB, Thomas-White KJ, Richter HE, Nager CW, Visco AG, Nygaard IE, Barber MD, Schaffer J, Moalli P, Sung VW, Smith AL, Rogers R, Nolen TL, Wallace D, Meikle SF, Gai X, Wolfe AJ, Brubaker L; Pelvic Floor Disorders Network. The female urinary microbiome in urgency urinary incontinence. Am J Obstet Gynecol. 2015 Sep;213(3):347.e1-11. doi: 10.1016/j.ajog.2015.07.009. Epub 2015 Jul 23. PMID 26210757
- [Background] Thomas-White KJ, Hilt EE, Fok C, Pearce MM, Mueller ER, Kliethermes S, Jacobs K, Zilliox MJ, Brincat C, Price TK, Kuffel G, Schreckenberger P, Gai X, Brubaker L, Wolfe AJ. Incontinence medication response relates to the female urinary microbiota. Int Urogynecol J. 2016 May;27(5):723-33. doi: 10.1007/s00192-015-2847-x. Epub 2015 Sep 30. PMID 26423260

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care Anticholinergic Treatment: Women presenting to the Urogynecology clinic with urgency urinary incontinence symptoms will receive standard of care anticholinergic treatment and will have their urinary microbiome evaluated before and after treatment
  Oxybutynin, Solifenacin, Tolterodine, Sanctura or Toviaz: Study participants will be evaluated for urgency urinary incontinence and will be offered treatment with a standard of care anticholinergic medication for 6 weeks. All study participants will fill out the UDI-6 and two day bladder diary at baseline before starting anticholinergic medication treatment. Participants will then provide a urine sample and blood draw to be assessed for urinary microbiome and inflammation. Anticholinergic medication will be taken daily for 6 weeks and the same procedures (UDI-6 questionnaire, bladder diary, urine sample except the blood draw for assessment) will be performed at the 6-week time period.
Period: Overall Study
Arm/Group | Standard of Care Anticholinergic Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Standard of Care Anticholinergic Treatment
Number analyzed (Participants) | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [52.5 to 73.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 20
Menopausal Status [Count of Participants; unit: Participants]
  Post-menopausal | 17
  Pre-menopausal | 3
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 0
  Past-smoker | 8
  Never-smoker | 12
Alcohol Use [Count of Participants; unit: Participants]
  Alcohol use | 11
  No alcohol use | 9
Caffeine Use [Count of Participants; unit: Participants]
  Caffeine use | 17
  No caffeine use | 3
HRT/Vaginal Estrogen Use [Count of Participants; unit: Participants]
  Hormone Replacement Therapy (HRT)/Vaginal Estrogen Use | 4
  No HRT/Vaginal Estrogen Use | 16
Contraceptive Use [Count of Participants; unit: Participants]
  Current contraceptive use | 2
  No contraceptive use | 18
Comorbidities [Count of Participants; unit: Participants]
  None | 11
  Diabetes | 4
  Heart disease | 1
  Hypertension | 8
  Stroke | 1
  Asthma/COPD | 4
  Depression/anxiety | 6
  Arthritis | 3
  Thyroid Disease | 2
  Liver Disease | 0
  Renal Disease | 0

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Markers in Urine Will be Measured Using Immunoenzyme Assays to Measure the Interaction of Anticholinergic Treatment and the Inflammatory Milieu.
Description: Statistical testing was used to determine if there was a difference in inflammatory markers in the urine of patients between baseline visit and 6 week visit. 7 markers were chosen and compared, all inflammatory markers present in urine.
Time Frame: Baseline and 6 weeks
Population: 20 patients were involved in the study, however only 13 returned for follow-up, hence 13 patients involved in "follow-up" group.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Anticholinergic Treatment
Number analyzed (Participants) | 20
pg/mL
  Baseline CRP | 2.192 [1.902 to 2.867]
  Follow-up CRP: number analyzed (Participants) | 13
  Follow-up CRP | 2.565 [1.900 to 3.758]
  Baseline IL-12/IL-23p40 | 2.192 [1.902 to 2.867]
  Follow-up IL-12/IL-23p40 | 2.565 [1.900 to 3.758]
  Baseline MCP-1 | 75.49 [55.69 to 117.85]
  Follow-up MCP-1 | 65.02 [37 to 109.79]
  Baseline GM-CSF | 0.102 [0.06 to 0.122]
  Follow-up GM CSF | 0.203 [0.092 to 0.272]
  Baseline IL-1B | 0.203 [0.106 to 0.542]
  Follow-up IL-1B | 0.415 [0.130 to 42.11]
  Baseline IL-6 | 0.667 [0.502 to 1.641]
  Follow-up IL-6 | 0.967 [0.749 to 2.951]
  Baseline IL-8 | 7.211 [4.85 to 23.044]
  Follow-up IL-8 | 6.116 [3.363 to 24.11]
Statistical Analysis 1: Comparison: Standard of Care Anticholinergic Treatment; T-test of Wilcoxon rank sum was used to test this non-normal data. Null hypothesis is that the concentration of urine inflammatory markers is the same at baseline and follow-up. This p-value is the probability that the difference in the CRP Calc. Conc. (pg/ml) between baseline and follow-up; Test type: Superiority; p = 0.6497, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Standard of Care Anticholinergic Treatment; T-test of Wilcoxon rank sum was used to test this non-normal data. Null hypothesis is that the concentration of urine inflammatory markers is the same at baseline and follow-up. This p-value is the probability that the difference in the IL-12/IL-23p40 Calc. Conc. (pg/ml) between baseline and follow-up; Test type: Superiority; p = 0.4281, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Standard of Care Anticholinergic Treatment; The null hypothesis is that the baseline and follow-up levels of the urine inflammatory markers are due to chance. This p-value represents the probability that the difference between the baseline and follow-up levels of MCP-1 Calc. Conc. (pg/ml) is due to chance; Test type: Superiority; p = 0.3157, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Standard of Care Anticholinergic Treatment; This p-value represents the probability that the difference between baseline and follow-up levels of GM-CSF Calc. Conc. (pg/ml) is due to chance; Test type: Superiority; p = 0.1463, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Standard of Care Anticholinergic Treatment; The null hypothesis is that the baseline and follow-up levels of the urine inflammatory markers are due to chance. This p-value represents the probability that the difference between the baseline and follow-up levels of IL-1β Calc. Conc. (pg/ml) is due to chance; Test type: Superiority; p = 0.6091, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Standard of Care Anticholinergic Treatment; The null hypothesis is that the baseline and follow-up levels of the urine inflammatory markers are due to chance. This p-value represents the probability that the difference between the baseline and follow-up levels of IL-6 Calc. Conc. (pg/ml) is due to chance; Test type: Superiority; p = 0.3011, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Standard of Care Anticholinergic Treatment; The null hypothesis is that the baseline and follow-up levels of the urine inflammatory markers are due to chance. This p-value represents the probability that the difference between the baseline and follow-up levels of IL-8 Calc. Conc. (pg/ml) is due to chance; Test type: Superiority; p = 0.5009, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: The Effectiveness of Anticholinergic Treatment in Relation to the Urinary Microbiome. Culture to Standard Culture Media Will Pickup Aerobic Bacteria and Yeasts After DNA Extraction and End Point PCR for 16S rDNA Genes.
Description: The change in g_lactobacillus from Baseline to Follow-up (6 weeks), which corresponds to before and after anticholinergic treatment.
Time Frame: At the 6 week mark
Population: The median change in g_lactobacillus for patients who had both baseline and follow-up samples analyzed.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Anticholinergic Treatment
Number analyzed (Participants) | 13
pg/mL | 0.001131599 [-0.020078049 to 0.102829877]

3. Secondary Outcome: The Urogenital Distress Inventory (UDI-6) Questionnaire Will be Used to Assess Baseline Urinary Symptoms Prior to Anticholinergic Treatment. Participants Indicate How Long They Have Had These Symptoms.
Description: Symptoms taken from the UDI-6, a validated questionnaire for urogynecologic symptoms, were gathered at baseline for all patients. Duration of Urinary Incontinence symptoms is presented.
Time Frame: Baseline visit (0 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Anticholinergic Treatment
Number analyzed (Participants) | 20
Participants
  <6 months | 8
  6-23 monts | 7
  2-4 years | 4
  5-10 years | 0
  >10 years | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of any patient being involved in the study. Since no patients were involved for more than 1 year, data was collected for 1 year total to ensure any and all adverse event data were caught.
Description: Our definition of adverse event did not differ.
Arm/Group | Standard of Care Anticholinergic Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04090190/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/90/NCT04090190/SAP_003.pdf